CLINICAL TRIAL: NCT03282084
Title: A Prospective, Observational Study of the PPI Non-responder
Status: Withdrawn | Type: Observational
Why Stopped: insufficient funding
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: D17109
Record Dates: First submitted 2017-06-09; First posted 2017-09-13 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Gastro Esophageal Reflux Disease PPI Non-Responders
MeSH Terms: interventions — Endoscopy, Digestive System; Biopsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unproven GERD: Subjects with no prior testing, normal prior EGD or prior LA Grade A esophagitis
  Interventions: Diagnostic Test: EGD with biopsy
- Proven GERD: LA Grade B-D esophagitis, long-segment Barrett's, prior positive pH study
  Interventions: Diagnostic Test: EGD and impedance-pH study on PPI

INTERVENTIONS:
Diagnostic Test: EGD with biopsy — Stop PPI and schedule for EGD with biopsy and Wireless pH capsule testing for 7-10 days later. Consider gastric emptying scan or high resolution esophageal manometry
  Other Names: Wireless pH Capsule
  Groups: Unproven GERD
Diagnostic Test: EGD and impedance-pH study on PPI — Continue PPI and schedule EGD and Impedance-pH study on PPI. Consider gastric emptying scan or high resolution esophageal manometry
  Groups: Proven GERD

SUMMARY:
Gastroesophageal reflux disease (GERD) is a common chronic condition, affecting approximately 20% of the American adult population. Proton pump inhibitors (PPIs) are now the mainstay of medical therapy for symptoms of GERD. Despite their efficacy, several studies have shown that a significant proportion of GERD patients are either partial or non-responders to PPI therapy, defined as symptoms of heartburn and/or regurgitation not relieved by either a standard or double dose of a PPI during a minimum trial of 8 weeks. If GERD symptoms persist, further testing is required. This study will mirror the real world setting to assess the value of published guidelines which recommend specific testing and treatment.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a common chronic condition, affecting approximately 20% of the American adult population. Gastroesophageal reflux disease is characterized by a number of symptoms, the 2 most common being frequent heartburn and acid regurgitation. Untreated or undertreated gastroesophageal reflux (GER) can lead to complications including esophageal erosions, strictures, esophageal adenocarcinoma, and impaired quality of life.

Proton pump inhibitors (PPIs) are now the mainstay of medical therapy for symptoms of GERD. Despite their efficacy, several studies have shown that a significant proportion of GERD patients are either partial or non-responders to PPI therapy, defined as symptoms of heartburn and/or regurgitation not relieved by either a standard or double dose of a PPI during a minimum trial of 8 weeks. A review of 19 studies looking at GERD patients treated with PPIs found an overall prevalence of partial and non-responders of up to 45% in observational studies. Non-randomized studies revealed a prevalence of 17% when defined as "persisting troublesome heartburn" and 28% when defined as troublesome regurgitation, while randomized studies revealed prevalence rates of 32% and 28%, respectively.

Current guidelines recommend an 8-week trial of a daily PPI for the treatment of symptoms thought secondary to GERD. However, if GERD symptoms persist despite taking the PPI correctly, then testing is required. National guidelines recommend that patients with GERD symptoms who have failed empiric therapy with a PPI undergo upper endoscopy (EGD). This recommendation is based on data showing that the PPI non-responsive patient may have a disorder (e.g., peptic ulcer disease, dyspepsia, eosinophilic esophagitis, cancer) that can only be identified by EGD. During upper endoscopy a 48-hour wireless pH capsule can be placed to measure acid reflux into the distal esophagus. This recommended practice has been shown to be cost effective. If the 48 hour wireless pH capsule study documents pathologic acid reflux, then the diagnosis of acid reflux is confirmed and the patient should be restarted on a PPI with appropriate counseling regarding how to take a PPI properly. Switching the patient to an alternative PPI is a reasonable strategy, as some patients respond better to one PPI than another . In addition, during this index endoscopy, biopsies of the esophagus should be taken to rule out eosinophilic esophagitis.

Some patients in clinical practice have previously undergone testing due to their GERD symptoms. In patients with proven GERD (e.g., prior EGD with LA Grade B-D esophagitis, known Barrett's esophagus, prior positive pH tests either on or off PPI therapy) who continue to have GERD symptoms on a daily PPI, guidelines recommend that impedance pH-testing be performed on daily PPI therapy. Guidelines do not recommend testing on b.i.d. PPI therapy, since most patients with GERD do not require twice-daily PPI therapy. In this patient population (the PPI non-responder with proven GERD), impedance-pH testing is preferable to 48-hour wireless pH capsule testing as non-acid reflux can be detected as well. To be cost effective, and to reduce the number of unnecessary EGDs, if upper endoscopy was recently performed, then impedance-pH testing can be performed after accurate localization of the lower esophageal sphincter using high resolution esophageal manometry (HREM). If the impedance-pH test is negative (normal) on daily PPI therapy, demonstrating that acid reflux is controlled, then a second diagnosis should to be considered (e.g., functional dyspepsia, gastroparesis, an esophageal motility disorder). If impedance-pH monitoring demonstrates abnormal acid reflux on daily PPI therapy, then guidelines recommend that the PPI dose should be increased to twice daily and symptoms reassessed at 8 weeks.

The clinical treatment pathways outlined above are based on national guidelines and are promoted as standards of care. However, despite the fact that these guidelines recommend distinct diagnostic pathways for patients who are non-responsive to PPIs, there is little "real-world" data to support these guidelines and no information about the outcomes of these patients who are treated using these diagnostic pathways. The simple goal of this study is to identify the PPI non-responder patient with GERD symptoms and identify and quantify the type, number and outcomes of diagnostic tests recommended by national guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign informed consent
* Persistent GERD symptoms after minimum 8 week trial on daily PPI

Exclusion Criteria:

* Unwilling to sign informed consent
* Prior anti-reflux surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent GERD symptoms despite treatment with a minimum of 8 weeks daily PPI.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Objectively evaluate PPI non-responder | 8 Weeks after visit 2
  Number of participants with unproven GERD who have reflux esophagitis and eosinophile esophagitis
Esophageal acid exposure | 8 Weeks after visit 2
  Number and extent of abnormal acid exposure as measured by pH-metry (Bravo capsule) off PPI.
Response to different PPI | 8 Weeks after visit 2
  Percentage of patients with GERD who fail standard PPI Therapy as documented by wireless pH capsule testing that then respond to an alternative PPI
Document the amount of esophageal acid and non-acid exposure in the PPI non-responder patient with proven GERD | 8 Weeks after visit 2
  Amount of acid and non-acid exposure in PPI-nonresponder patients with proven GERD as measured by impedance-pH testing on daily PPI therapy.
Determine the type, frequency and extent of esophageal motility disorders | 8 Weeks after visit 2
  Determine the type, frequency and extent of esophageal motility disorders using HREM (high resolution esophageal manometry) in patients with persistent GERD symptoms despite PPI therapy
Nepean Dyspepsia Index | 8 Weeks after visit 2
  Using a validated questionnaire determine the prevalence and severity of functional dyspepsia in patients presenting with GERD symptoms using the Nepean Dyspepsia Index.
Correlate subjective symptoms of GERD with objective evidence of acid reflux | 8 Weeks after visit 2
  Comparison of symptomatic GERD based on GERD-Q validated questionnaire and pH testing
Assess overlapping symptoms of dysphagia and GERD | 8 Weeks after visit 2
  Assess overlapping symptoms of dysphagia in patients with GERD symptoms who do not respond to empiric PPI therapy using a validated dysphagia questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Lacy, MD, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Locke GR 3rd, Talley NJ, Fett SL, Zinsmeister AR, Melton LJ 3rd. Prevalence and clinical spectrum of gastroesophageal reflux: a population-based study in Olmsted County, Minnesota. Gastroenterology. 1997 May;112(5):1448-56. doi: 10.1016/s0016-5085(97)70025-8. PMID 9136821
- [Background] Nebel OT, Fornes MF, Castell DO. Symptomatic gastroesophageal reflux: incidence and precipitating factors. Am J Dig Dis. 1976 Nov;21(11):953-6. doi: 10.1007/BF01071906. PMID 984016
- [Background] El-Serag H, Becher A, Jones R. Systematic review: persistent reflux symptoms on proton pump inhibitor therapy in primary care and community studies. Aliment Pharmacol Ther. 2010 Sep;32(6):720-37. doi: 10.1111/j.1365-2036.2010.04406.x. PMID 20662774
- [Background] Richter JE. How to manage refractory GERD. Nat Clin Pract Gastroenterol Hepatol. 2007 Dec;4(12):658-64. doi: 10.1038/ncpgasthep0979. PMID 18043675
- [Background] Cicala M, Emerenziani S, Guarino MP, Ribolsi M. Proton pump inhibitor resistance, the real challenge in gastro-esophageal reflux disease. World J Gastroenterol. 2013 Oct 21;19(39):6529-35. doi: 10.3748/wjg.v19.i39.6529. PMID 24151377
- [Background] Katz PO, Gerson LB, Vela MF. Guidelines for the diagnosis and management of gastroesophageal reflux disease. Am J Gastroenterol. 2013 Mar;108(3):308-28; quiz 329. doi: 10.1038/ajg.2012.444. Epub 2013 Feb 19. No abstract available. PMID 23419381
- [Background] Dickman R, Boaz M, Aizic S, Beniashvili Z, Fass R, Niv Y. Comparison of clinical characteristics of patients with gastroesophageal reflux disease who failed proton pump inhibitor therapy versus those who fully responded. J Neurogastroenterol Motil. 2011 Oct;17(4):387-94. doi: 10.5056/jnm.2011.17.4.387. Epub 2011 Oct 31. PMID 22148108
- [Background] Lee WC, Yeh YC, Lacy BE, Pandolfino JE, Brill JV, Weinstein ML, Carlson AM, Williams MJ, Wittek MR, Pashos CL. Timely confirmation of gastro-esophageal reflux disease via pH monitoring: estimating budget impact on managed care organizations. Curr Med Res Opin. 2008 May;24(5):1317-27. doi: 10.1185/030079908x280680. Epub 2008 Mar 27. PMID 18377705
- [Background] Miller SM, Goldstein JL, Gerson LB. Cost-effectiveness model of endoscopic biopsy for eosinophilic esophagitis in patients with refractory GERD. Am J Gastroenterol. 2011 Aug;106(8):1439-45. doi: 10.1038/ajg.2011.94. Epub 2011 Mar 29. PMID 21448144
- [Background] Charbel S, Khandwala F, Vaezi MF. The role of esophageal pH monitoring in symptomatic patients on PPI therapy. Am J Gastroenterol. 2005 Feb;100(2):283-9. doi: 10.1111/j.1572-0241.2005.41210.x. PMID 15667483
- [Background] Mainie I, Tutuian R, Shay S, Vela M, Zhang X, Sifrim D, Castell DO. Acid and non-acid reflux in patients with persistent symptoms despite acid suppressive therapy: a multicentre study using combined ambulatory impedance-pH monitoring. Gut. 2006 Oct;55(10):1398-402. doi: 10.1136/gut.2005.087668. Epub 2006 Mar 23. PMID 16556669
- [Background] Quigley EM, Lacy BE. Overlap of functional dyspepsia and GERD--diagnostic and treatment implications. Nat Rev Gastroenterol Hepatol. 2013 Mar;10(3):175-86. doi: 10.1038/nrgastro.2012.253. Epub 2013 Jan 8. PMID 23296247
- [Background] Camilleri M, Parkman HP, Shafi MA, Abell TL, Gerson L; American College of Gastroenterology. Clinical guideline: management of gastroparesis. Am J Gastroenterol. 2013 Jan;108(1):18-37; quiz 38. doi: 10.1038/ajg.2012.373. Epub 2012 Nov 13. PMID 23147521